CLINICAL TRIAL: NCT04667676
Title: Respiratory Functions Response To Tens Acupoint Stimulation Post Inhalation Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-12-2020
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Inhalation Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS Therapy Group (Experimental): patients received acupoint TENS
  Interventions: Device: acupoint TENS
- Control group (Sham Comparator): patients received shame acupoint TENS
  Interventions: Device: acupoint TENS

INTERVENTIONS:
Device: acupoint TENS — TENS was applied bilaterally on acupoint Ex-B1, 4Hz frequency, and 200 μs pulse width and intensity was set at the best highest tolerable intensity by the patient sensitivity without a sensation of discomfort for 45 minutes, three times/week for four weeks

SUMMARY:
this study designed to examine the effect of Acu-TENS applied bilaterally on Ding Chuan acupoint to boost pulmonary functions, improve diaphragmatic excursion and decrease dyspnea in patients with inhalation injuries.

ELIGIBILITY:
Inclusion Criteria:

* Partial or full-thickness major burns
* Diagnosis of smoke inhalation based on the history of smoke exposure and chest computed tomography (CT)
* Have no systemic disease
* Body mass index less than 30.

Exclusion Criteria:

* Patients with any other pulmonary condition
* Cardiac condition
* Rib fracture
* Systemic disease
* Local infection and cigarette or tobacco use

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Spirometer | 4 weeks
  • Portable spirometer to measure forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) from setting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt